CLINICAL TRIAL: NCT05025501
Title: Family Based Executive Function Training for Schoolage Children With ADHD - A Randomized Controlled Study
Brief Title: A Randomized Controlled Study of Family Based EF Training for Schoolage Children With ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: XH-21-006
Record Dates: First submitted 2021-08-25; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: ADHD; Child, Only
Keywords: ADHD; executive function; schoolage; family-based intervention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects in this group will receive the "Famliy based Executive Function Training " program in aiming to reduce ADHD symptoms and improve the executive function.
  Interventions: Behavioral: Family based Executive Function Training
- Waiting group (No Intervention): Subjects in this group will not receive the "Famliy based Executive Function Training " program during the study period.

INTERVENTIONS:
Behavioral: Family based Executive Function Training — Training the executive funtions of shcoolage ADHD children through tasks and games repeatly but with fun. Giving the parental training and support for the parenting role parents strategies to help the shcoolage ADHD childred coping the symptoms and develop EF in the reallife and improve parent-child relationship.
  Arms: Intervention group

SUMMARY:
The goal of this study is to provide a new treatment approach for schoolage children with ADHD, which could facilitate the EF developing well to achieve better outcome.

DETAILED DESCRIPTION:
ADHD in preschoolers has become established as a valid psychiatric disorder with characterized core deficits of executive function (EF). The EF impairments occurred in preschool period could persist to childhood, adolescent and adulthood, causing extensive and deep damage of individual's academic and career achievement, social function, and peer relationship. Although medication showed significant effectiveness in controlling the core symptoms of ADHD, it failed to help patients master compensatory strategies to cope with functional impairments in learning and life events. The family intervention program for school-age ADHD children is still rare, and it is a blank field in China. At present, most of these related studies have not integrated task training in realistic scenarios with parent training, and lack of randomized and controlled Settings, which makes the effect of intervention less convincing. Therefore, the investigators conduct this randomized and controlled study to find out the therapeutic efficacy of Family-based Executive Function Training for Schoolage Children with ADHD, and follow the subjects to observe whether the therapeutic efficacy would persist. In the mean time, the investigators also observe the factors which can influence the therapeutic efficacy. The goal of this study is to provide a new treatment approach for schoolage children with ADHD, which could facilitate the EF developing well to achieve better outcome.

ELIGIBILITY:
Inclusion Criteria:

1. meet both the criteria of ADHD based on the interview by the CDIS and clinical diagnosis with DSM-5;
2. full-scale IQ estimated bythe Wechsler Intelligence Scale for Children-Revised Form (WISC-R) above 80;
3. their parents volunteered to participate in this study.

Exclusion Criteria:

1. child with severe mental disorder or physical disease that might interfere the assessment and intervention, such as Autistic Spectrum Disorder(ASD), Schizophrenia, epilepsy, traumatic brain injury, etc.;
2. parents with severe mental illness, such as schizophrenia, mood disorder (period of onset), etc..

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-06 (Estimated); Study Completion 2022-02-06 (Estimated)

PRIMARY OUTCOMES:
The executive function of of schoolage child of ADHD | through the intervention completion, an average of 12 weeks
  The core symptoms of schoolage children of ADHD assessed by neuropsychological evaluation tool NEPSY

SECONDARY OUTCOMES:
The executive function in real life of schoolage child of ADHD | through the intervention completion, an average of 12 weeks
  The executive function in real life of schoolage children of ADHD assessed by BRIEF
The ADHD symptoms of child | through the intervention completion, an average of 12 weeks
  The ADHD symptoms of child assessed by SNAP

CONTACTS AND LOCATIONS:
Overall Officials: Meihui Qiu, Master, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided